CLINICAL TRIAL: NCT03181412
Title: Evaluation of the Performances of the Cincinnati Prehospital Stroke Severity Scale Realized During Telephone Call With Emergency Department Physicians to Predict Large-vessel Occlusion
Brief Title: Stroke Cincinnati Prehospital Stroke Severity Scale Evaluation iN prEhospital
Acronym: SCENE
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0146
Record Dates: First submitted 2017-06-07; First posted 2017-06-08 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Pain Measurement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with suspected ischemic stroke: The cohort will be constituted of patients treated for a stroke suspicion after calling emergency medical services of the Rhone and presenting a symptom-onset (the last time the patient was seen without deficit) less than 6 hours.
  Interventions: Diagnostic Test: Questionnaire

INTERVENTIONS:
Diagnostic Test: Questionnaire — Tests from Cincinnati prehospital stroke severity scale (CPSSS) will be carried out by the physician at emergency medical services on telephone call with firemen, paramedics or the emergency medical services team for any stroke suspicion that meets the criteria for inclusion. Emergency department physician will have to follow a standardized questionnaire to complete the different items of the score. The score will not be calculated by emergency department physician and will not influence the orientation and management of patients.
  The final diagnosis will be the presence or absence of a large vessel occlusion. This diagnosis will be done on cerebral imaging by a neurologist.

SUMMARY:
The effectiveness of acute ischemic stroke (AIS) management has improved considerably in recent years with thrombolysis and more recently with mechanical thrombectomy (MT). Currently, mechanical thrombectomy can only be performed in stroke unit with an interventional neuroradiology center by experienced/qualified interventional neuroradiologists. In the Rhone area, only one hospital has the authorization to perform mechanical thrombectomy. Therefore, transferring directly eligible acute ischemic stroke patients for mechanical thrombectomy to this center constitutes an important stake of the triage of suspected acute ischemic stroke patients. Some validated scores for the identification of severe strokes and large vessel occlusion, including the Cincinnati prehospital stroke severity scale (CPSSS), appear to be relevant for pre-hospital use in order to identify patients potentially eligible for mechanical thrombectomy and address them to a stoke unit with interventional radiology center.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients calling emergency medical services for suspected acute ischemic stroke

Exclusion Criteria:

* Symptom onset (or the last time the patient was seen without deficit ) of more than 6 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stroke of the Rhone area after emergency medical services call
Sampling Method: Non-Probability Sample
Enrollment: 1272 (Actual)
Dates: Start 2018-06-25 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Performances of Cincinnati prehospital stroke severity scale | 1 day
  The Cincinnati prehospital stroke severity scale is composed of 3 items: 2 points if the patient has a deviation of the gaze, 1 point if the patient is not able to give the date and answer to a simple order such as closing the eyes or clenching the fist and 1 point if the patient presents a hemiplegia. The CPSSS score ranges from 0 to 4, highest value indicating the worst score. It will be considered positive if it is equal to 2 or more.
  Performances will be evaluated in terms of sensitivity, specificity, positive and negative predictive values.

CONTACTS AND LOCATIONS:
Locations (12):
- France (12):
  - Neurologie, Hôpital Neurologique - HCL, Bron
  - SAMU 69 , Hôpital Edouard Herriot, Lyon
  - Médecine d'urgence, Clinique de la Sauvegarde, Lyon
  - Médecine d'urgence, Hôpital de la Croix-Rousse - HCL, Lyon
  - Médecine d'urgence, Hôpital Desgenettes, Lyon
  - Médecine d'urgence, Hôpital Mutualiste Médipôle, Lyon
  - Médecine d'urgence, Hôpital Saint Joseph Saint Luc, Lyon
  - Urgentiste, Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Médecine d'urgence, CH de Roanne, Roanne
  - Médecine d'urgence, Hôpital Nord-Ouest, Tarare
  - Services Médecine d'urgence et Neurologie, CH de Vienne, Vienne
  - Services Neurologie et Médecine d'urgence, CH de Villefranche sur Saône, Villefranche-sur-Saône

IPD SHARING:
Plan to Share IPD: No